CLINICAL TRIAL: NCT05481931
Title: Non-Interventional Post-Authorisation Safety Study of NUCEIVA for the Treatment of Moderate-to-Severe Glabellar Lines
Brief Title: Non Interventional Safety Study of NUCEIVA for the Treatment of Moderate-to-Severe Glabellar Lines
Status: Active, not recruiting | Type: Observational
Sponsor: Evolus, Inc. (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Other Study IDs: EV-010
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — prabotulinumtoxin A

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (3):
- Safety Population: The safety population will consist of all patients who receive at least one treatment of NUCEIVA.
  Interventions: Drug: prabotulinumtoxinA
- Botulinum Toxin Naïve: Sub-population of patients that have never been treated with botulinum toxin
  Interventions: Drug: prabotulinumtoxinA
- Botulinum Toxin Exposed: Sub-population of patients that have previously been treated with botulinum toxin
  Interventions: Drug: prabotulinumtoxinA

INTERVENTIONS:
Drug: prabotulinumtoxinA — Botulinum toxin Type A powder for solution for injection
  Other Names: Jeuveau; Nuceiva

SUMMARY:
Non-interventional PASS of NUCEIVA for the treatment of moderate-to-severe glabellar lines to provide additional characterisation of the long-term safety of NUCEIVA in the real-world clinical practice setting.

DETAILED DESCRIPTION:
This is a prospective, multicentre, non-interventional observational Post Authorisation Safety Study; Safety data will be collected from approximately 750 patients at 20 sites throughout the United Kingdom and the European Union over an 18 month evaluation period. Eligible patients will receive an initial treatment of 20 Units of NUCEIVA. Further treatment will not be specified, recommended or required by the protocol. Patients may receive up to 6 treatments of 20 Units of NUCEIVA over the course of the 18-month study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is an adult less than 65 years of age
* Patient presenting to a participating physician has moderate to severe vertical lines between the eyebrows seen at maximum frown (glabellar lines)
* Patient finds their glabellar lines have an important psychological impact
* Written informed consent is obtained from the patient.

Exclusion Criteria:

* Patient has a legal incapacity or limited legal capacity without legal guardian representation
* Patient is currently participating in an interventional study of any investigational product, device or procedure
* Patient has a hypersensitivity to the active substance or to any of the excipients listed in Section 6.1 of the Summary of Product Characteristics
* Patient has a generalised disorder of muscle activity (e.g. myasthenia gravis or Eaton Lambert Syndrome)
* Patient has an infection or inflammation at any of the proposed injection sites
* Patient has a history of dysphagia and/or aspiration
* Female patient is pregnant, is of childbearing potential and not using contraception, is breast feeding, or is planning to become pregnant during the next 18 months
* Patient has received prior botulinum toxin for any indication within 3 months of study enrolment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Approximately 750 patients will be recruited at 20 sites from the United Kingdom, Germany, France, Sweden and Spain.
Sampling Method: Probability Sample
Enrollment: 756 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events | From the time of first dose until participant exits the study at 18 months post initial treatment
  Number and percentage of patients with an event that started or worsened in severity at or after the first dose of NUCEIVA

SECONDARY OUTCOMES:
Adverse Events of Particular Interest | From the time of first dose until participant exits the study at 18 months post initial treatment
  Number and percentage of patients that experience an adverse event related to eye disorders and adverse events potentially suggestive of the distant spread of toxin.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Avelar, Study Director — Evolus, Inc.
Locations (1):
- Cologne Dermatology, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No